CLINICAL TRIAL: NCT00646971
Title: Exhaled Markers of Oxidative Stress and Endothelium-dependent Vascular Relaxation in Obstructive Sleep Apnea. Effect of Continuous Positive Airway Pressure Therapy.
Brief Title: Oxidative Stress and Endothelial Dysfunction in Obstructive Sleep Apnea
Acronym: SOREVAS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insuffisent recrutment
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Mathieu QUINTIN, Departement Clinical Research of Developpement
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P041012
Record Dates: First submitted 2008-03-17; First posted 2008-03-31 (Estimated); Last update posted 2010-07-12 (Estimated); Status verified 2010-05

CONDITIONS: Obstructive Sleep Apnea Syndrome; Endothelial Dysfunction; Oxidative Stress; Intermittent Hypoxia; Cardiovascular Risk
Keywords: Isoprostane; Alkane; Exhaled condensate; Peripheral arterial tonometry; Polysomnography; Obstructive Sleep Apnea; Hypoxia
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypoxia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): CPAP
  Interventions: Device: CPAP device
- 2 (Sham Comparator): sham CPAP
  Interventions: Device: Placebo device

INTERVENTIONS:
Device: CPAP device — for 4 weeks
  Other Names: CPAP
  Arms: 1
Device: Placebo device — for 4 weeks
  Other Names: Placebo
  Arms: 2

SUMMARY:
Patients with sleep apnea syndrome have repeated apneic events that induce periodic hypoxia-reoxygenation, drawing away an overproduction of oxidants. This exaggerated generation of oxidants is associated with a dysfunction of the vascular endothelium that evolves, in its turn, towards cardiovascular diseases such as systemic hypertension, stroke, and myocardial infarction. The major aim of our study is to examine the effect of CPAP treatment on biochemical (markers of oxidative stress) and functional (endothelium-dependent vascular relaxation reactivity) abnormalities at 1 and 4 weeks of treatment.

DETAILED DESCRIPTION:
Subjects will undergo overnight polysomnography in the sleep laboratory (PSG1, D0), which will be immediately preceded and followed by measurements of oxidative stress in exhaled gas and vascular relaxation. Patients included in the OSAS group will be randomly assigned to treatment by either CPAP or Placebo (sham CPAP) for 4 weeks. Measurements of oxidative stress in exhaled gas and vascular reactivity will be repeated immediately before and after PSG2 and PSG3 at D7 and D30, respectively.

ELIGIBILITY:
Inclusion Criteria:

* No smoking
* 30-70 years old subjects
* being referred for daytime hyper- somnolence and snoring
* apnea hypopnea index >=30/hour and desaturation index>=30/hour

Exclusion Criteria:

* Chronic lung diseases.
* Exposure to occupational contaminants.
* Active smoking within last 2 years.
* Alcoholism.
* Chronic systemic disease other than OSAS.
* Treatment with vasoactive drugs or antioxidants
* Respiratory infection or vaccination during the 6 weeks preceding the PSG1.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
To examine the effect of CPAP treatment on biochemical (markers of oxidative stress) abnormalities | 1 and 4 weeks of treatment

SECONDARY OUTCOMES:
To compare between patients with severe OSAS and controls, the degree of the production of markers of oxidative stress non-invasively measured in both the exhaled gas and urine samples | before and after a nocturnal polysomnography
To compare between patients and controls, the endothelium-dependent vascular relaxation | before and after nocturnal polysomnography
To analyze the relationship between these biochemical and functional abnormalities and the standard criteria of severity of OSAS. | before and after nocturnal polysomnography
To examine the effect of CPAP treatment on functional (endothelium-dependent vascular relaxation reactivity) abnormalities | 1 and 4 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pierre ESCOURROU, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris Hôpital Antoine Béclère; Gabriel ROISMAN, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris, Hôpital Antoine Béclère
Locations (1):
- Assistance Publique - Hôpitaux de Paris Hôpital Antoine Béclère, Clamart, France